CLINICAL TRIAL: NCT06872138
Title: S100A8 in Serum and Urine as a New Biomarker in Lupus Nephritis
Status: Completed | Type: Observational
Sponsor: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Ghada Khalifa Sayed, Assistant Professor of Nephrology, Theodor Bilharz Research Institute (TBRI), Giza, Egypt, Theodor Bilharz Research Institute
Other Study IDs: PT(882)
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: S100A8; Serum; Urine; Biomarker; Lupus; Nephritis
MeSH Terms: conditions — Nephritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Systemic lupus erythematosus (SLE) Group: Systemic lupus erythematosus (SLE) patients.
  Group I will be subdivided into two groups:
  Group IA (n=30): SLE patients with lupus nephritis (LN) Group IB (n=20): SLE patients without LN.
- Control Group: Age and sex matched healthy control

SUMMARY:
This study aims to evaluate both serum and urine S100A8 as potential biomarkers for Lupus nephritis (LN)

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a systemic autoimmune/ inflammatory disease that can affect any organ of the human body. The molecular pathophysiology of SLE remains largely unknown, but complex interactions of genetic factors, the environment, and hormones contribute to disease expression.

Clinical importance of S100 calcium-binding protein A8 protein (S100A8) as a biomarker in SLE has been well-established. During an inflammatory reaction, neutrophils produce S100A8, a Ca2+-binding protein that is part of the S100 family and is found in neutrophil extracellular traps.

In addition to its primary role as a member of the S100A8/A9 heterodimer, S100A8 accumulates in various bodily compartments and functions as a damage-associated molecular pattern molecule upon release. It is a crucial regulator of inflammation and enhances the function of innate immune cells by interacting with members of the immunoglobulin superfamily of cell surface molecules, such as toll-like receptor 4 and the receptor of advanced glycation end products.

Serum S100A8 levels are linked with disease activity, glomerulonephritis, and anti-double-stranded DNA (dsDNA) antibodies (Ab), according to increasing experimental and clinical data. healthy controls (HCs) had lower serum S100A8 levels. Considering that elevated blood S100A8 levels are also seen in several inflammatory disorders such as inflammatory bowel disease and rheumatoid arthritis, it is unclear if this elevated level is adequate to serve as a biomarker specific to SLE.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* Patients with Systemic lupus erythematosus (SLE)
* Patients with SLE and renal affection. SLE diagnosis is based on the 1997 American College of Rheumatology (ACR) criteria or the 2012 Systemic Lupus International Collaborating Clinics (SLICC) classification criteria.

Renal involvement (lupus Nephritis) (LN) can be diagnosed by presence of proteinurea or elevated kidney function and can be confirmed by biopsy if present.

Exclusion Criteria:

* Autoimmune diseases.
* Sjogren's syndrome.
* Rheumatoid arthritis.
* Systemic sclerosis.
* Taking other biologic disease-modifying anti-rheumatic drugs.
* Immunosuppressive drugs.
* Corticosteroid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants were stratified into two main groups: Group I consisted of 50 SLE patients, further subdivided into Group IA (n=30) with LN and Group IB (n=20) without LN. Group II comprised 20 age- and sex-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-03-30 (Actual)

PRIMARY OUTCOMES:
Assessment of S100A8 levels in serum for diagnosing lupus nephritis (LN) | 3 months
  Venous blood (5cm blood) and urine will be collected from patients with systemic lupus erythematosus (SLE) and healthy control, and the serum will be immediately centrifuged at 15,928 relative centrifugal force (RCF) and for 10 min. The supernatant will be collected and stored at -80°C until further analysis.
  Before the enzyme-linked immunosorbent assay (ELISA) is conducted, frozen serum samples will be thawed and then diluted 1:100 in phosphate-buffered saline. S100A8 homodimer concentrations will be measured using a commercially available ELISA kit for serum.

SECONDARY OUTCOMES:
Accessment S100A8 levels in urine for diagnosing lupus nephritis (LN) | 3 months
  Venous blood (5cm blood) and urine will be collected from patients with systemic lupus erythematosus (SLE) and healthy control, and the serum will be immediately centrifuged at 15,928 relative centrifugal force (RCF) and for 10 min. The supernatant will be collected and stored at -80°C until further analysis.
  Before the enzyme-linked immunosorbent assay (ELISA) is conducted, frozen urine samples will be thawed and then diluted 1:100 in phosphate-buffered saline. S100A8 homodimer concentrations will be measured using a commercially available ELISA kit for urine.
Correlation between S100A8 level and disease activity markers | 3 months
  Correlation between S100A8 level and disease activity markers in patients with systemic lupus erythematosus will be measured
Using S100A8 as a predictor for renal affection in systemic lupus erythematosus (SLE) patients for follow up and early treatment. | 3 months
  Renal involvement lupus Nephritis can be diagnosed by presence of proteinurea or elevated kidney function and can be confirmed by biopsy if present.

CONTACTS AND LOCATIONS:
Locations (1):
- Theodor Bilharz Research Institute, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding autho